CLINICAL TRIAL: NCT05581823
Title: A Phase 1, Open-label, Fixed-sequence, Crossover Trial to Evaluate the Effects of Cytochrome P450 (CYP) 3A4 Induction by Carbamazepine on the Steady-state Pharmacokinetics of Tavapadon in Healthy Adult Participants
Brief Title: Study to Evaluate the Effects of Cytochrome P450 (CYP) 3A4 Inducer Carbamazepine on Tavapadon Pharmacokinetics in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-751-1005
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tavapadon Followed by Tavapadon + Carbamazepine (Experimental): Participants will receive oral tavapadon tablets titrated up to a steady-state dose from Day 1 to Day 14. From Day 15, participants will receive oral carbamazepine tablets titrated up to a steady-state dose along with oral tavapadon tablets, up to Day 30.
  Interventions: Drug: Tavapadon; Drug: Carbamazepine

INTERVENTIONS:
Drug: Tavapadon — Oral tablets
  Other Names: CVL-751; PF-06649751
Drug: Carbamazepine — Extended-release oral tablets

SUMMARY:
The primary purpose of this study is to evaluate the effect of carbamazepine, a strong CYP3A4 inducer, on the steady-state pharmacokinetics (PK) of tavapadon in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Women of nonchildbearing potential and men 18 to 55 years, inclusive, at the time of signing the informed consent form (ICF).
2. Sexually active men with a pregnant or nonpregnant partner of childbearing potential must agree to use a condom during the trial and for 90 days after the last dose of carbamazepine. In addition, male participants should not donate sperm for a minimum of 90 days following the last dose of carbamazepine.
3. Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator.
4. Body mass index of 18.5 to 32.0 kilograms per square meter (kg/m^2), inclusive, and total body weight >50 kg (110 pounds [lbs]) at Screening.
5. Capable of giving signed informed consent as described in the full protocol, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
6. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. "Yes" responses for any of the following items on the C-SSRS (within past 6 months):

   * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
   * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) "Yes" responses for any of the following items on the C-SSRS (within past 2 years):
   * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior).

   Serious risk of suicide in the opinion of the investigator is also exclusionary.
2. Participants shown to carry or be positive for human leukocyte antigen (HLA)-B*1502 or HLA-A*3101.
3. Use of prohibited medication prior to randomization (5 half-lives) or likely to require prohibited concomitant therapy (e.g., prescription and over-the-counter medications, herbal medications, vitamins, and supplements) during the trial. CYP3A4 inhibitors and inducers are prohibited from 30 days prior to signing of the ICF through the end of the trial.
4. Recent monoamine oxidase inhibitors (MAO-I) use (in the last 28 days) as it increases the risk for hypersensitivity and bone marrow suppression from carbamazepine.
5. Prior carbamazepine use that was discontinued for tolerability or adverse events, including a clinically significant decrease in platelets, white blood cells or hemoglobin.
6. Platelets, white blood cell count, or hemoglobin <lower limit of normal (LLN).
7. Estimated glomerular filtration rate <90 milliliters per minute (mL/min)/1.73 m^2, as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

NOTE: Other protocol-defined Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 31
Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCτ) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 31

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and AEs by Severity | Day 1 up to Day 36
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to Day 31
Number of Participants with Clinically Significant Changes in Vital Sign Values | Up to Day 31
Number of Participants with Clinically Significant Changes in Clinical Laboratory Assessments | Up to Day 30
Number of Participants with Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 31
Changes in Suicidality Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Day 31
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Madison, Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No